CLINICAL TRIAL: NCT01676259
Title: A Prospective, Multinational, Multi-Center, Phase 2, Single-Arm, Open-Label Study Evaluating the Efficacy, Safety and Tolerability of siG12D-LODER in Combination With Standard of Care Chemotherapy in the Treatment of Patients With Locally Advanced Pancreatic Cancer
Brief Title: A Phase 2 Study of siG12D LODER in Combination With Chemotherapy in Patients With Locally Advanced Pancreatic Cancer
Acronym: PROTACT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Silenseed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLSG12D-P2
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
Keywords: siRNA; RNA interference (RNAi); Cancer; Pancreatic ductal adenocarcinoma; Locally Advanced Pancreatic cancer; Solid tumor; Non operable pancreatic ductal adenocarcinoma; Borderline resectable
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Drug Therapy; folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- siG12D-LODER + chemotherapy (Experimental): Eight siG12D-LODER+Gemcitabine+nab-Paclitaxel or Eight siG12D-LODER+Folfirinox or Eight siG12D-LODER+modifide Folfirinox
  Interventions: Drug: siG12D-LODER; Drug: Gemcitabine+nab-Paclitaxel; Drug: Folfirinox

INTERVENTIONS:
Drug: siG12D-LODER — The implantation of siG12D-LODERs is selected to meet current gastroenterology endoscopic ultrasound (EUS) biopsy procedures, proved to be highly effective and safe.
Drug: Gemcitabine+nab-Paclitaxel — Gemcitabine+nab-Paclitaxel
  Other Names: Chemotherapy
Drug: Folfirinox — Folfirinox or modified Folfirinox
  Other Names: Chemotherapy

SUMMARY:
In this Phase II study a dose of 2.8 mg (eight 0.35 mg siG12D-LODERs) will be administered in 12-week cycles to patients with unresectable or borderline resectable locally advanced pancreatic cancer combined with chemotherapy treatment.

Primary Outcome:

- ORR at 6 months.

DETAILED DESCRIPTION:
In this Phase II study a dose of 2.8 mg (eight 0.35 mg siG12D-LODERs) will be administered in 12-week cycles to patients with unresectable or borderline resectable LAPC combined with chemotherapy treatment (Gemcitabine+nab-Paclitaxel or Folfirinox or modified Folfirinox). This will be a study to assess the response rate of the siG12D-LODER in patients with unresectable or borderline resectable LAPC. The study is of a single arm design with one arm receiving siG12D-LODER + chemotherapy.

The investigational agent siG12D-LODER is a miniature biodegradable bio polymeric matrix that encompasses the drug, designed and produced by Silenseed Ltd. The implantation of LODERs is selected to meet current gastroenterology endoscopic ultrasound (EUS) biopsy procedures, proved to be highly effective and safe.

siG12D-LODER has been studied in the escalating dose Phase I study of 15 patients, and results showed high safety and tolerability profiles, with no single DLT.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Subject must be 18 years of age or older at the time of signing the informed consent.

Type of Subject and Disease Characteristics

1. Histologically or cytologically confirmed adenocarcinoma of the pancreas.
2. Locally advanced pancreatic cancer stage III according to The American Joint Committee on Cancer (AJCC) and defined as T4, N (any) and M0, according to the three factors, T (tumor), N (node involvement), and M (metastases), of the National Comprehensive Cancer Network TNM classification.
3. Allocated to receive one of the following chemotherapies: gemcitabine plus nab-paclitaxel, FOLFIRINOX or modified FOLFIRIONOX as first line treatment for pancreatic cancer.
4. Have a target tumor that is accessible for intratumoral administration by EUS as determined by the radiologist/gastroenterologist performing the EUS intratumoral administration, according to The American Society for Gastrointestinal Endoscopy (ASGE) guidelines (https://www.asge.org/home/practice-support/guidelines).
5. Have measurable disease. Subject will have a histologically-confirmed disease and must have clinically and/or radiographically documented measurable primary disease according to RECIST v1.1. At least one site of disease must be unidimensionally measurable.

   Diagnostic Assessments
6. Eastern Cooperative Oncology Group (ECOG) Performance Scale of ≤ 1.
7. Demonstrate adequate organ function as defined below:

   * serum creatinine <1.6 mg/dL
   * international normalized ratio (INR) < 1.5 U
   * absolute neutrophil count (ANC) > 1.5 x 109/L
   * platelets ≥ 100 x 109/L
   * hemoglobin ≥ 9 mg/dL
   * alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 5 times upper limit of normal (ULN)
   * bilirubin ≤ 1.5 x ULN Sex
8. Male and/or female. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
9. Women of childbearing potential (WOCBP): a negative serum or urine pregnancy test during screening.
10. Subject of childbearing potential, if sexually active (both men and women) must agree to use a barrier method of contraception, from the time of administration of the first treatment and for at least 8 weeks after EOT visit day.

    Informed Consent
11. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Subjects with resectable pancreatic cancer.
2. Evidence of metastatic disease.
3. Other malignancy that would interfere with the current intervention.
4. Any evidence of ascites (beyond trace).
5. Bulky celiac adenopathy (≥2.5 cm) or non-adenocarcinoma histology.
6. Previously treated malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancers from which the subject has been disease-free for at least 2 years.
7. History of clinically significant coagulopathy.
8. Major surgery, other than diagnostic surgery, within 4 weeks prior to study entry without complete recovery.
9. New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 4 months prior to the first chemotherapy cycle Day 1, unstable arrhythmia or symptomatic peripheral arterial vascular disease.
10. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
11. Known active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus.
12. Females who are pregnant or breast-feeding.
13. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.

    Prior/Concomitant Therapy
14. Any prior therapy for the treatment of pancreatic malignancy (including chemotherapy, immunotherapy, vaccines, monoclonal antibodies, major surgery, or irradiation, whether conventional or investigational).
15. Prior therapy with any hypoxic cytotoxic agent (hypoxia-targeting drugs). Prior/Concurrent Clinical Study Experience
16. Subjects who are participating or participated in an investigational drug or device study (within 28 days prior to study entry from the last study dose date).

    Other Exclusions:
17. Unwillingness or inability to comply with the study protocol for any reason.
18. Known allergy to sesame oil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
ORR at 6 months | One year

CONTACTS AND LOCATIONS:
Overall Officials: Eileen M O'Reilly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Talia Golan, MD, Principal Investigator — Sheba Medical Center
Locations (9):
- United States (4):
  - Hackensack Meridian Health, Hackensack, New Jersey
  - The Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Israel (5):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center (Tel H'shomer), Ramat Gan
  - Sourasky MC (Ichilov) Tel Aviv Israel, Tel Aviv
  - Assaf Harofeh Medical Center, Tzrifin